CLINICAL TRIAL: NCT02784977
Title: TURKAPNE - The Turkish Sleep Apnea Database: A National, Multicenter, Observational, Prospective Cohort Study
Acronym: TURKAPNE
Status: Recruiting | Type: Observational
Sponsor: Koç University (Other)
Collaborators: Ege University School of Medicine, Izmir, Turkey (Unknown); Dokuz Eylul University (Other); Diskapi Yildirim Beyazit Education and Research Hospital (Other Government); Uludag University (Other); Dicle University School of Medicine, Diyarbakir, Turkey (Unknown); Namik Kemal University School of Medicine, Tekirdag (Other); Suleyman Demirel University School of Medicine, Isparta, Turkey (Unknown); Istanbul University - Cerrahpasa (Other); Pamukkale University School of Medicine, Denizli, Turkey (Unknown); Trakya University (Other); Afyon Kocatepe University School of Medicine, Afyon, Turkey (Unknown); Hitit University School of Medicine, Corum, Turkey (Unknown); Istanbul Sureyyapasa Chest Diseases and Chest Surgery Training and Research Hospital (Other); Kocaeli Education and Research Hospital, Kocaeli, Turkey (Unknown); Baskent University Ankara Hospital (Other); Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2016.311
Record Dates: First submitted 2016-05-18; First posted 2016-05-27 (Estimated); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Conservative Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Obstructive Sleep Apnea (OSA): Patients with apnea hypopnea index of at least 5 events per hour. Intervention with positive airway pressure, or intraoral device, or uvuloplasty, or conservative treatment.
  Interventions: Device: Positive Airway Pressure (PAP); Device: Intraoral device (IOD); Procedure: Uvuloplasty; Other: Conservative treatment
- No-OSA: Patients with apnea hypopnea index less than 5 events per hour. No intervention.

INTERVENTIONS:
Device: Positive Airway Pressure (PAP) — Treatment of OSA with PAP
  Groups: Obstructive Sleep Apnea (OSA)
Device: Intraoral device (IOD) — Treatment of OSA with IOD
  Groups: Obstructive Sleep Apnea (OSA)
Procedure: Uvuloplasty — Uvuloplasty
  Groups: Obstructive Sleep Apnea (OSA)
Other: Conservative treatment — No active intervention
  Groups: Obstructive Sleep Apnea (OSA)

SUMMARY:
Primary aim of the TURKAPNE (The Turkish Sleep Apnea Database) study is to generate a cross-sectional nationwide database to define clinical and polysomnographic characteristics of the sleep apnea patients in Turkey. Associations of phenotypes of sleep apnea patients with metabolic and cardiovascular diseases as well as risk for traffic accidents will be explored as secondary aims. Impact of treatment of sleep apnea on metabolic and cardiovascular complications as well as compliance with positive airway pressure treatment will be further explored longitudinally.

DETAILED DESCRIPTION:
All subjects undergoing sleep study for suspicion of obstructive sleep apnea will be registered in a web-based national database regarding:

* Anthropometric data, educational status, driving licence,
* Smoking and alcohol use
* Comorbidities, and drug use
* Questionnaires, excessive daytime sleepiness
* Polygraphic and polysomnographic findings
* Blood pressure measurements
* If taken, blood glucose, lipids and other biochemical markers
* If measured, lung function test results
* If measured, echocardiography findings
* Follow-up data regarding treatment modality and compliance

ELIGIBILITY:
Inclusion Criteria:

* Consecutive adult patients undergoing sleep study for suspicion of obstructive sleep apnea
* Ability to read and speak
* Signed informed consent.

Exclusion Criteria:

* subjects who use positive airway pressure
* subjects with limited life expectancy due to advanced renal disease or uncontrolled malignancies
* subjects with alcohol dependency

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients referred to the sleep clinics for suspicion of sleep apnea
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2017-10-03 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Metabolic and cardiovascular diseases in obstructive sleep apnea phenotypes | Up to three years
  The association of sleep apnea severity indices such as Apnea-Hypopnea Index and Oxygen Desaturation Index during Rapid Eye Movement (REM) sleep and non-REM sleep with self-reported diabetes mellitus and cardiovascular diseases will be explored.

SECONDARY OUTCOMES:
Sex differences in obstructive sleep apnea phenotypes | Up to three years
  Possible sex differences in REM-dependent sleep apnea, positional sleep apnea and its association with metabolic and cardiovascular diseases will be explored
Adherence to positive airway pressure treatment in obstructive sleep apnea | Through study completion, an average of 7 years
  Predictors of adherence to positive airway pressure treatment (defined as device usage at least 4 hours of night during at least 70% of study period) in obstructive sleep apnea
Incidence of cardiovascular diseases and mortality | Through study completion, an average of 7 years
  Number of patients who have died or developed cardiovascular diseases

CONTACTS AND LOCATIONS:
Overall Officials: Yüksel Peker, Prof, Study Chair — Koç University School of Medicine, Dept of Pulmonary Medicine; Özen Kacmaz Basoglu, Prof, Principal Investigator — Ege University School of Medicine; Hikmet Firat, Assoc. Prof, Principal Investigator — Ankara Diskapi Yildirim Beyazit Education and Research Hospital; Oya Itil, Prof, Principal Investigator — Dokuz Eylul University Medical School; Mehmet Karadag, Prof, Principal Investigator — Uludag University Medical School; Nejat Altintas, Assoc. Prof, Principal Investigator — Namik Kemal University Medical School; Gökhan Kirbas, Prof, Principal Investigator — Dicle University Medical School; Önder Öztürk, Assoc. Prof, Principal Investigator — Süleyman Demirel University Medical School; Derya Karadeniz, Prof, Principal Investigator — Istanbul University Cerrahpasa Medical School; Nese Dursunoglu, Assoc. Prof, Principal Investigator — Pamukkale University Medical School; Gundeniz Altiay, Prof, Principal Investigator — Trakya University Medical School; Ersin Günay, Assoc. Prof, Principal Investigator — Afyon Kocatepe University Medical School; Sema Sarac, MD, Principal Investigator — Istanbul Sureyyapasa Education and Research Hospital; Zahide Yilmaz, MD, Principal Investigator — Kocaeli Education and Research Hospital; Aylin Ozsancak Ugurlu, Assoc. Prof, Principal Investigator — Istanbul Baskent University Hospital; Kadriye Agan Yildirim, Prof, Principal Investigator — Marmara University, Faculty of Medicine, Department of Neurology; Sertac Arslan, Assist Prof, Principal Investigator — Corum Hitit University
Locations (1):
- Koç University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peker Y, Basoglu OK, Firat H; TURKAPNE Study Group. Rationale and Design of the Turkish Sleep Apnea Database - TURKAPNE: A National, Multicenter, Observational, Prospective Cohort Study. Turk Thorac J. 2018 Jul;19(3):136-140. doi: 10.5152/TurkThoracJ.2018.18097. Epub 2018 Jul 1. PMID 30083405
- [Derived] Pihtili A, Kiyan E, Balcan B, Arbatli S, Cilli A, Altintas N, Ugurlu AO, Gurkan CG, Tasbakan MS, Dursunoglu N, Ogun H, Annakkaya AN, Sokucu SN, Firat H, Basoglu OK, Peker Y; Turkapne Study Group. Sex differences in clinical and polysomnographic features of obstructive sleep apnea: The Turkish sleep apnea database (TURKAPNE) cohort. Sleep Med. 2025 Feb;126:228-234. doi: 10.1016/j.sleep.2024.12.018. Epub 2024 Dec 17. PMID 39721358